CLINICAL TRIAL: NCT01599845
Title: The Differential Pattern of Deposition of Nano Particles in the Airways of Exposed Workers (Nanoexposure)
Brief Title: The Differential Pattern of Deposition of Nano Particles in the Airways of Exposed Workers
Acronym: Nanoexposure
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-11-YS-0107-CTIL
Record Dates: First submitted 2012-04-29; First posted 2012-05-16 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Inadequate or Impaired Respiratory Function
Keywords: Lung; Alveoli; Nanoparticles; Particulate matter; Exhaled breath condensate; Induced sputum; Forced expiratory volume; Force vital capacity
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nanoparticle exposed

SUMMARY:
Investigation of the differences between the levels of extracellular and intracellular nano-particles in workers exposed to environmental particles during their employment to enhance understanding the process of penetration of the particles to respiratory epithelial cells.

DETAILED DESCRIPTION:
This study investigates the following questions:

Does occupational exposure to nanoparticles influence permeation of such particles to respiratory airways? Is there a correlation between the levels of nanoparticles in sample biological fluids of the patients and their pulmonary functions.

Is there a correlation between the levels of nanoparticles in sample biological fluids of the patients and respiratory tract infections.

The study protocol includes the following steps:

Initial interview of the patient Measurement of nanoparticles in samples of exhaled breath condensate using NanoSight LM 20 Measurement of nanoparticles in induced sputum. And finally examination of the relationship between the measured parameters and the indices of pulmonary infection, and pulmonary function as measured by the pulmonary department of the TASMC.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years of age who visit Ichilov Hospital for medical complaints/inquiries regarding respiratory tract.
* Study population is composed of people who are exposed to environmental particles form industrial sources.
* Informed consent is requested from each subject.

Exclusion Criteria:

* Unemployed individuals.
* Individuals who are not working in industrial jobs, such as office workers and secretaries.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Analysis of the size distribution of nano-particles in exhaled breath condensate | One year
  Each subject will be examined once. The total time for collection of data is estimated as about one year.

CONTACTS AND LOCATIONS:
Overall Officials: Yehuda Schwarz, M.D., Principal Investigator — Tel Aviv Sourasky Medical Center (TASMC, Ichilov)